CLINICAL TRIAL: NCT06595056
Title: Primary Care Referrals to a Remotely Delivered Physical Activity Intervention for Latina Teens: Chicas Fuertes 2
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Family Health Centers of San Diego (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Britta Larsen, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 810268; R01HL171807 (NIH)
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-05

CONDITIONS: Physical Activity
Keywords: adolescent health; Latina; teenager; mHealth; fitness tracker
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will receive a one-on-one counseling session and access to an individually tailored multi-media website. Key intervention components will be reinforced through text messaging to aid goal setting, a physical activity tracker (Fitbit) to set goals, track and log activity, and access to a study Instagram account to reinforce exposure to web content.
  Interventions: Behavioral: Multi-technology MVPA intervention
- Control (No Intervention): Participants will receive a physical activity tracker (Fitbit) only.

INTERVENTIONS:
Behavioral: Multi-technology MVPA intervention — Participants will receive a one-on-one counseling session and access to an individually tailored multi-media website. Key intervention components will be reinforced through text messaging to aid goal setting, a physical activity tracker (Fitbit) to set goals, track and log activity, and access to a study Instagram account to reinforce exposure to web content.
  Arms: Intervention

SUMMARY:
This study will test a physical activity intervention for Latina teenagers. Investigators will recruit 200 Latina adolescents who are currently under-active to participate in this 12-month study. Participants will be referred to the study by their primary care provider. Half of the participants will be randomly selected for the Intervention group, and will receive an individual counseling session and access to a personalized website. These participants will also receive a Fitbit activity tracker to help with goal setting and monitoring, plus weekly text messages and access to the study Instagram account to remind participants to be physically active. Those assigned to the control group will receive the Fitbit activity tracker.

DETAILED DESCRIPTION:
This study will conduct a randomized trial to evaluate the efficacy of a theory-based, individually tailored, multi-technology intervention on increasing physical activity in Latina adolescents, compared to a control group receiving only a physical activity tracker (a Fitbit). The study team will recruit adolescent (age 13-17) Latinas (N=200) who are currently under-active to participate in the 12-month trial. Those randomized to the Intervention arm will receive a one-on-one counseling session and access to an individually tailored multi-media website. Key intervention components will be reinforced through text messaging to aid goal setting, a physical activity tracker (Fitbit) to set goals, track and log activity, and access to a study Instagram account to reinforce exposure to web content. The primary outcome will be increases in moderate-to-vigorous activity between baseline and 6 months. Secondary outcomes will include changes in activity at 12 months, potential mediators of the intervention, costs of delivering the intervention, behavior change trajectories from continuous data from Fitbits, potential moderators, and changes in physiological and psychological variables.

ELIGIBILITY:
Inclusion Criteria:

* self identify as Latina
* age 13-17
* read, write, and speak English
* be a current patient at FHCSD
* be under-active (engaging in 60 min/day of MVPA on fewer than 5 days per week)
* regular access (≥2 times/week) to Internet and a smart phone that can receive text messages

Exclusion Criteria:

* unwillingness to be randomized to one of the two conditions
* self-reporting any condition that would impair ability to participate in physical activity for at least 10 minutes at a time

Ages: 13 Years to 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Meeting guidelines for physical activity | 6 months
  Proportion of participants meeting guidelines of 60 min/day of moderate to vigorous physical activity (MVPA) measured by Fitbits

SECONDARY OUTCOMES:
Maintenance of MVPA | 12 months
  Proportion of participants meeting guidelines of 60 minutes/day of MVPA measured by Fitbits.
Processes of Change for Physical Activity (POC) | 12 months
  Questionnaire that tracks cognitive and behavioral processes related to MVPA change
Stages of Change for Physical Activity (SCPA) | 12 months
  Questionnaire that determines what stage of exercise engagement the participant is currently in (precontemplation, contemplation, preparation, action, maintenance), and is used to stage-match treatment.
Self-Efficacy for Physical Activity (SE) | 12 months
  Questionnaire that measures self-efficacy to become physically active across diverse contexts
Social Support for Exercise (SSE) | 12 months
  Questionnaire measuring social support specifically in relation to exercise with three subscales (friends, family, rewards/punishments)
Outcome Expectations Scale | 12 months
  Questionnaire that measures the beliefs regarding the consequences of physical activity participation
Technology Engagment | 12 months
  Tracks activity on the study website (logins, goal setting, questionnaires answered), Fitbit activity (days worn, sync frequency), texting activity (% of interactive texts responded to), Instagram activity (views, likes)
Neighborhood Environment Walkability Scale for Youth (NEWS-Y) | Baseline
  Questionnaire that measures perceptions of neighborhood environment including recreation facility availability, pedestrian traffic safety, and walking facilities
Vital Signs | 12 months
  Height, weight, resting blood pressure
Perceived Stress Scale (PSS) | 12 months
  Questionnaire used to assess stress levels
Demographics | Baseline
  Age, race, parent education and income, marital status, acculturation
Physical Activity Enjoyment Scale (PACES) | 12 months
  Questionnaire that assesses level of personal satisfaction from physical activity
Childrens Depression Inventory (CDI) | 12 months
  Questionnaire that measures affective, cognitive, motivational, and somatic symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- University of California- San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All quantitative data produced in the course of the project will be preserved and shared. Transcripts from stakeholder interviews will be shared only in the event that they give permission for the entire transcript to be shared; otherwise, summaries and codebooks will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Shared data generated from this project will be made available as soon as possible, and no later than the time of publication or the end of the funding period, whichever comes first. The duration of preservation and sharing of the data will be a minimum of 7 years after the end of the funding period.
Access Criteria: The Larsen USCD data provides metadata, persistent identifiers and long-term access. This repository is supported by USCD and dataset(s) are available through a request process directly with the PI, Dr. Larsen.

REFERENCES:
- [Background] Larsen B, Greenstadt ED, Olesen BL, Marcus BH, Godino J, Zive MM. An mHealth Physical Activity Intervention for Latina Adolescents: Iterative Design of the Chicas Fuertes Study. JMIR Form Res. 2021 Jun 15;5(6):e26195. doi: 10.2196/26195. PMID 34128823